CLINICAL TRIAL: NCT03901222
Title: 3D Analysis of the Effects of tDCS on a Functional Task in High Level Athletes
Brief Title: 3D Analysis of the Effects of tDCS (Transcranial Direct Current Stimulation) on a Functional Task in High Level Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Bornheim Stephen, Assistant Professor, University of Liege
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 2017/309
Record Dates: First submitted 2019-03-28; First posted 2019-04-03 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Healthy; Athlete
Keywords: tDCS; Athlete; Endurance; Fatigue; 3D
MeSH Terms: conditions — Fatigue | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Randomized, triple-blind, sham-controlled, crossover
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The device is preprogrammed by a third party non participating in any element in the study. They then chose (using opaque envelopes) the treatment code for each participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bi-Anodal tDCS (Active Comparator): Subjects will receive 20 min of bi-anodal tDCS
  Interventions: Device: tDCS
- Sham tDCS (Sham Comparator): Subjects will receive 20 minutes of Sham anodal tDCS
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — 20 minutes of anodal tDCS (C3 & C4/FPZ) 2mA or sham
  Other Names: Non invasive brain stimulation

SUMMARY:
Relatively high level athletes will undergo 2 randomized, cross-over counterbalanced sessions of bi-anodal tDCS (transcranial direct current stimulation) or sham tDCS The primary outcome is a 3D evaluation coupled with EMG (Electromyography) of their primary lower limb muscles after each session

DETAILED DESCRIPTION:
Recruitment :

Relatively high level athletes will be recruited through social media and advertisements.

Each subject came twice to the Liege University Hospitals' Human Movement Analysis Laboratory.

After placing the different infrared emitters and placing and calibrating the surface EMG electrodes, subjects underwent 3 maximal squat jumps (without upper limb implication). They were then familiarized with the fatigue protocol (8 jumps at a 33 jumps per minute pace).

Then each subject received either bi-anodal tDCS of sham tDCS. Neither the evaluator or the subject knew which they were receiving. Immediately following tDCS, subjects underwent another warmup 3 maximal squat jumps, and then the fatigue protocol (comprised of 30 maximal jumps at a rate of 33 per minute).

ELIGIBILITY:
Inclusion Criteria:

* At least 10 hours of sport a week
* Right handed and footed

Exclusion Criteria:

* One on the TSST (in high and relatively high risk sections)
* Previous neurological or orthopedic pathologies affecting limbs

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-03-31 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Peak Height | Changes between Prior and Immediately Following tDCS and Sham
  Peak height (measured by the 3D device) is measured after each of the 30 repetitions as well as after the 3 jumps before and after tDCS. Height decrease will also be looked at
Gluteal EMG (Electromyography) recordings (% of maximal EMG value) | Changes between Prior and Immediately Following tDCS and Sham
  Bilateral Gluteal EMG
Quadriceps EMG (Electromyography) recordings (% of maximal EMG value) | Changes between Prior and Immediately Following tDCS and Sham
  Bilateral Quadriceps EMG triceps surae will be measured
Triceps EMG (Electromyography) recordings (% of maximal EMG value) | Changes between Prior and Immediately Following tDCS and Sham
  Bilateral Triceps Surae EMG

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Bornheim, Msc, Principal Investigator — Liege University Hospital
Locations (1):
- Liege Univeristy Hospital, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No